CLINICAL TRIAL: NCT05462236
Title: A Phase II Open Label, Dose-finding run-in and Cohort Expansion Study to Evaluate the Safety, Tolerability and Effectiveness of Tinodasertib in Combination With Pembrolizumab or Irinotecan in Metastatic Colorectal Cancer
Brief Title: MNK Inhibitor AUM001 in Combination With Either Pembrolizumab or Irinotecan to Treat Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AUM Biosciences Pte Ltd (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUM001-2001-MK3475-D65; KEYNOTE-D65 (Other: Merck Sharpe & Dohme Corp.); MK-3475-D65 (Other: Merck Sharpe & Dohme Corp.)
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Module 1: Arm A: Multiple dose finding cohorts (Experimental): Monotherapy with Tinodasertib administered orally QOD
  Interventions: Drug: Tinodasertib
- Module1: Arm B/C: Multiple cohorts of Tinodasertib with fixed dose of pembrolizumab or irinotecan (Experimental): Combination doses with Tinodasertib administered orally QOD with intravenous pembrolizumab at 200mg Q3W or Irinotecan at 180mg/m2 Q2W
  Interventions: Drug: Tinodasertib; Drug: Pembrolizumab; Drug: Irinotecan
- Module 2: Arm B' and C': Dose Expansion (Experimental): Combination therapy with Tinodasertib administered orally QOD at RP2D (as determined in Module 1) and either pembrolizumab at 200mg IV Q3W (arm B') or irinotecan 180mg/m2 IV Q2W (arm C')
  Interventions: Drug: Tinodasertib; Drug: Pembrolizumab; Drug: Irinotecan

INTERVENTIONS:
Drug: Tinodasertib — MNK inhibitor
  Other Names: AUM001
Drug: Pembrolizumab — PD-1 Inhibitor
  Other Names: KEYNOTE-D65; KEYTRUDA®
  Arms: Module 2: Arm B' and C': Dose Expansion; Module1: Arm B/C: Multiple cohorts of Tinodasertib with fixed dose of pembrolizumab or irinotecan
Drug: Irinotecan — Topoisomerase inhibitor
  Arms: Module 2: Arm B' and C': Dose Expansion; Module1: Arm B/C: Multiple cohorts of Tinodasertib with fixed dose of pembrolizumab or irinotecan

SUMMARY:
The study is a 2-part study of Tinodasertib alone or in combination with Pembrolizumab/Irinotecan in patients with CRC.

DETAILED DESCRIPTION:
The study is conducted in 2 parts. First a dose escalation Run-in to identify the Maximum Tolerable Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of Tinodasertib to be administered orally as monotherapy and in combination with intravenous pembrolizumab/irinotecan. Part 2 consists of a cohort expansion at the RP2D of Tinodasertib n combination with intravenous pembrolizumab/Irinotecan in patients with locally advanced or metastatic CRC to evaluate clinical activity and safety of Tinodasertib.

ELIGIBILITY:
Main Inclusion criteria:

1. The participant provides written informed consent for the trial.
2. Subjects are at least 18 years of age at the time of signing the Informed Consent Form
3. Subjects with histologically or cytologically confirmed diagnosis of locally advanced or metastatic CRC.

   1. Locally determined histological diagnosis is acceptable for study entry in Module 1.
   2. Subjects can be enrolled in module 1 regardless of microsatellite stability status.
   3. Only subjects with CRC MSS will be enrolled in module 2, arm B'.
4. Subjects who have had >2 lines of prior therapy for their CRC.

   1. Prior use of irinotecan or irinotecan containing regimens is permitted
   2. CRC MSI-H patients should have been treated with a checkpoint inhibitor and have progressed on such therapy or found to be resistant, refractory or intolerant to the checkpoint inhibitor
   3. Patients with an available molecularly targeted therapy such as antibodies targeting VEGF/R, EGFR, encorafenib/cetuximab, prior to study entry. Additionally, patients with driver mutations for which an FDA approved therapy is available such as BRAF V600E, HER2 or NTRK should have been offered such therapy prior to study entry.
   4. CRC subjects will be eligible to enrol in Arm C' if they have failed an established 5-fluorouracil containing regimen and have progressed after oxaliplatin based or irinotecan-based combination therapy and do not have a driver mutation for which there is an approved targeted therapy.
5. Subject must have provided archival tumor tissue sample or newly obtained core or excisional or punch needle biopsy of a tumor lesion not previously irradiated.
6. Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiologist.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
8. Have a predicted life expectancy of greater or equal to 3 months.
9. Have adequate organ function
10. HIV infected participants must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease
11. Women of childbearing potential must not be breastfeeding and must have a negative serum or urine pregnancy test. Must be willing to use an adequate method of contraception.
12. Women of non-childbearing potential: Evidence of post-menopausal status is required.
13. Male subjects: Non-sterilized male subjects who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide. Male subjects should refrain from sperm donation throughout this period.

Main Exclusion Criteria

1. Has a history of another malignancy within 2 years prior to first investigational product administration, unless the malignancy was treated with curative intent and the likelihood of relapse is <5% in 2 years.
2. Has known active CNS metastases and/or carcinomatous meningitis.
3. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives, whichever is shorter prior to study treatment.
4. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
5. Has had an allogeneic tissue/solid organ transplant.
6. Pregnant or breastfeeding
7. Has a known history or Hepatitis B (defined as HbsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
8. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
9. Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
10. Gastrointestinal (GI) tract disease causing the inability to take oral medication.
11. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor, and was discontinued from that treatment due to a Grade 3 or higher irAE.
12. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, or have had history of radiation pneumonitis.
13. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Adverse events and Serious Adverse events | Approximately 2 years from date of participant enrolment
  Incidence and severity of AEs and SAEs.
Incidence of DLT events and treatment emergent AEs (TEAEs) | 1 complete cycle (21 days)
  Grading of DLTs according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0
Objective response rate based on Response Evaluation Criteria in Solid tumors (RECIST) Version 1.1 | Approximately 2 years from date of participant enrolment

SECONDARY OUTCOMES:
PK evaluation | Approximately 6 months from date of participant enrolment
  Evaluation of Plasma concentrations of AUM001 as monotherapy or in combination with Pembrolizumab/Irinotecan

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Prince of Wales Hospital, Wollongong, New South Wales
  - Pindara Private Hospital, Gold Coast Cancer Care, Benowa, Queensland
  - Cabrini Hospital, Malvern, Victoria
  - Ballarat Oncology and Haematology, Wendouree, Victoria

IPD SHARING:
Plan to Share IPD: No